CLINICAL TRIAL: NCT06345651
Title: Brain Oscillation Synchronized Stimulation of the Frontal Cortex: Randomized Controlled Trial Comparing Frontal Theta-oscillation Synchronized Repetitive TMS With Standard TMS in Major Depressive Disorder
Brief Title: Brain Oscillation-synchronized Stimulation of the Frontal Cortex in Major Depressive Disorder
Acronym: BOSSFRONT2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-03, Version 7
Record Dates: First submitted 2024-01-08; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-01

CONDITIONS: Major Depressive Disorder
Keywords: Noninvasive Brain Stimulation; Transcranial magnetic stimulation; TMS; Personalized Medicine; Closed-Loop; Brain Oscillation; Depression; TBS
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: The study is a single-site randomized standard TMS therapy-controlled double-blind paral-lel-group design clinical trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In both conditions the identical setup is used consisting of Neuronavigation, EEG and TMS. Only in the experimental condition the treatment will be EEG-informed. In the control condition the treatment will be applied indepentently of the EEG signal.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Theta negative peak triggered TMS of left dmPFC (Experimental): Repetitive TMS (100 Hz triple pulses) of the dmPFC will be applied daily for four weeks (5 sessions per week on working days, 20 sessions in total). Stimulation triggers will be brain oscillation-synchronized based on EEG extracted over left dmPFC, synchronized with the negative peak of endogenous theta oscillations in left dmPFC.
  Interventions: Device: Transcranial Magnetic Stimulation
- iTBS TMS of left dlPFC (Active Comparator): Standard intermittent Theta Burst Stimulation of the dlPFC will be applied daily for four weeks (5 sessions per week on working days, 20 sessions in total). Stimulation triggers will be applied independently of the EEG signal.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Individually MR-neuronavigated TMS, 600 pulses, 120% RMT

SUMMARY:
Major depressive disorder (MDD) is a common severe psychiatric disease with enormous socioeconomic costs for the patient and society alike. Current pharmacological treatments are ineffective in a substantial fraction of patients and are accompanied by unwanted side effects. Using a novel non-invasive brain stimulation method to specifically target and modulate dysfunctional brain oscillations with high spatial and temporal precision this study will investigate the efficacy of EEG-triggered transcranial magnetic stimulation to alleviate de-pressive symptomatology in patients with MDD in a double-blind randomized controlled pilot clinical trial.

DETAILED DESCRIPTION:
Evidence from rTMS in the motor system suggests that synchronization of the individual TMS pulses with the negative (in a reference-free Laplacian transform) peak of endogenous EEG-derived brain oscillations results in LTP-like increase in cortical excitability, with the negative peak corresponding to a high-excitability state. A previous proof-of-principle study (BOSSFRONT, funded in the "AKF Anreizprogramm") showed that this approach can be used in patients suffering from major depressive disorder. Recent data from our lab in healthy volunteers indicates that the negative peak of frontocentral theta oscillations may play a similar role in frontal networks, and was therefore chosen with a dorsomedial prefrontal stimulation target in this study aiming to demonstrate therapeutic efficacy of a brain-oscillation synchronized stimulation protocol. The study is a single-site randomized standard TMS therapy-controlled double-blind parallel-group design clinical trial comparing theta-synchronized rTMS over left DMPFC with standard iTBS over left DLPFC in 30 patients with MDD. The primary outcome measure of the study is the difference in MADRS change (baseline / end of treatment) between the two treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have to be 18 to 65 years old
* Subjects meet DSM-5 criteria for current major depressive disorder (MDD), confirmed with the Structured Clinical Interview for DSM-5.
* Subjects score 20 points or more on the Montgomery-Åsberg Depression Rating Scale (MADRS).
* Subjects must have had at least one non-response (meaning a failure to achieve remission) in a previous pharmacological antidepressant treatment trial of sufficient (meaning a doses considered to be effective (e.g., superior to placebo in controlled clinical trials) and the duration needs to be sufficient to produce a ro-bust therapeutic effect (e.g., 12 weeks)) dosage and duration as assessed by the ATHF; treatment failure can be for the current or any prior depressive episode; medication resistance for the current episode is not required.
* Subject is in good physical and mental health. Subject understands the study procedures and agrees to participate in the study by giving written informed consent.
* Subject is willing to comply with the study restrictions.
* If antidepressant medication is being taken, it has to be taken for at least 2 weeks before inclusion in the study and the dose or active substance must not have been changed. It is necessary that no change in medication will be made until the end of the study (last visit takes place 4 weeks after the last therapy session). If a change in medication is necessary, further study participation is no longer possible.

Exclusion Criteria:

* Subject is under the age of legal consent.
* Subject has a diagnosis of bipolar disorder.
* Subject suffers from current symptoms of psychosis.
* Subject has active suicidal ideation with plan and/or intent.
* A current major depressive episode longer than 5 years.
* Subject has a history of substance abuse or dependence within the past 2 years.
* Subject has a diagnosis of antisocial or borderline personality disorder.
* Subject suffers from other major psychiatric or medical comorbidity
* Subject has a history of seizure disorder
* Subject has a history of severe head injury with loss of consciousness.
* Subject had a prior brain surgery
* Subjects with intake of pro-convulsive medication, e.g. imipramine, amitriptyline, doxepin, nortriptyline, maprotiline, chlorpromazine, clozapine, foscarnet, ganciclovir, ritonavir, amphetamines, cocaine, MDMA (ecstasy), phencyclidine (PCP, angel's dust), ketamine, gamma-hydroxybutyrate (GHB), alcohol, theophylline, in accord with present consensus guidelines on safety, ethical considerations, and application of TMS in clinical practice and research.
* Daily intake of Benzodiazepines other than Lorazepam >1 mg/d
* Subject has a cardiac pacemaker, implanted medication pump, intracardiac line, or acute, unstable cardiac disease.
* Subject has an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head (excluding the mouth) that cannot be safely removed.
* Subject has participated in another study within 2 weeks prior to the first study visit.
* Subject has contra-indications to MRI scans or does not agree that (1) the scans are obtained for research purposes only and will not be evaluated by a qualified neuroradiologist; if an abnormality is present, this may well not be noticed by the doctors, scientists and other staff involved in the study and handling the MRI da-ta; and that (2) if any of the staff involved in the study do suspect a relevant ab-normality to be present in any of the scans, they will reveal this to the subject so that a further diagnostic workup can be conducted outside of the study.
* Subject is pregnant or trying to get pregnant. If someone is not sure weather she is pregnant or not we will test HCG in the urine.
* Planned or anticipated changes of medication within the study period. If a change in medication is necessary, further study participation is no longer possible.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | baseline, immediately after the intervention
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is a questionnaire for external assessment of the severity of a depressive syndrome. The questionnaire consists of 10 questions. The questions are rated on a 7-point scale from 0 to 6. The total score ranges from 0 (best outcome) to 60 (worst outcome) points by summing up. The questionnaire is considered gold standard in the assessment of depressive symptoms. It will be performed at baseline and at the end of the treatment.

SECONDARY OUTCOMES:
MADRS (Montgomery-Åsberg Depression Rating Scale) 4 weeks after intervention | 4 weeks after the last interventional session
  Difference in MADRS change 4 weeks after the last treatment session vs. baseline measurement on the day of the first treatment session between the two treatment arms.
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is a questionnaire for external assessment of the severity of a depressive syndrome. The questionnaire consists of 10 questions. The questions are rated on a 7-point scale from 0 to 6. The total score can be between 0 (best outcome) and 60 (worst outcome) after summing up. The questionnaire is considered gold standard in the assessment of depressive symptoms. It will be performed at baseline and at the end of the treatment.
HDRS-17 (Hamilton Depression Rating Scale-17) | baseline, immediately after the intervention
  The HDRS-17 (Hamilton Depression Rating Scale-17) is designed to rate the severity of depression in patients. The rating is performed by a clinician. A score of 0-7 is considered to be normal while a score of 20 or higher indicates at least moderate severity.
BDI-2 (Beck Depression Inventory-2) | baseline, immediately after the intervention
  BDI-2 (Beck Depression Inventory-2) is a 21-question multiple-choice self-report inventory and represents the most widely used psychometric test for assessing the severity of depression in patients. 29-63 points reflect a severe depression.
IDS-30 (Inventory of depressive symptoms-30) | baseline, immediately after the intervention
  The IDS-30 (Inventory of depressive symptomes-30) is considered equivalent to or superior to the standard Hamilton Depression Scale (HAMD) and Beck Depression Inventory (BDI) tests. The scores ranges from 0 to 84 points.
  Patients with scores from 39 are considered severely depressed.
Response Rate | immediately after the intervention
  Response rate (50% reduction from MADRS) after the last treatment vs. measurement on the day of the first treatment session
Remission Rate | immediately after the intervention
  Remission rate (MADRS under 9 points) after the last treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Ziemann, Prof., Study Director — University Hospital Tuebingen; Andreas J Fallgatter, Prof., Study Director — University Hospital Tuebingen
Locations (1):
- University Hospital Tuebingen, Tübingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Lieb A, Zrenner B, Becker-Sadzio J, Gordon PC, Kozak G, Zrenner C, Martus P, Ziemann U, Fallgatter A. Brain oscillation-synchronized stimulation for major depression: a randomized controlled trial comparing EEG-triggered repetitive TMS with standard iTBS (Acronym: BOSSFRONT2). Eur Arch Psychiatry Clin Neurosci. 2026 Jan 21. doi: 10.1007/s00406-025-02176-9. Online ahead of print. No abstract available. PMID 41563436